CLINICAL TRIAL: NCT05524064
Title: FLASH Radiotherapy for the Treatment of Symptomatic Bone Metastases in the Thorax
Acronym: FAST-02
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Varian, a Siemens Healthineers Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VAR-2022-03
Record Dates: First submitted 2022-08-21; First posted 2022-09-01 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Bone Metastases in the Thorax
Keywords: FLASH radiotherapy; Radiation treatment; Proton; Bone metastasis; Pain relief; Toxicities; Thorax; Ultra-high dose rate

STUDY DESIGN:
Intervention Model Description: Open label, single arm prospective study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- FLASH radiotherapy for painful bone metastasis(-es) (Experimental): FLASH radiotherapy is radiation treatment delivered at ultra-high dose rates compared to conventional radiation treatment.
  Interventions: Radiation: FLASH Radiotherapy

INTERVENTIONS:
Radiation: FLASH Radiotherapy — A dose of 8 Gy delivered in a single fraction will be prescribed to the PTV, delivered with FLASH Radiotherapy (>40 Gy/s).

SUMMARY:
The purpose of this study is to assess toxicities of FLASH radiotherapy treatment and pain relief in subjects with painful thoracic bone metastases. FLASH radiotherapy is radiation treatment delivered at ultra-high dose rates compared to conventional radiation treatment.

DETAILED DESCRIPTION:
This clinical investigation is designed to assess the toxicities of FLASH radiotherapy treatment, as well as pain relief when used to treat bone metastasis(-es) in the thorax. Workflow metrics of FLASH radiotherapy in the thorax in a clinical setting will also be assessed. Patients at least 18 years of age with painful bone metastases located in the thorax will be considered for the study. Eligible subjects will be treated for painful bone metastases in the thorax using a palliative regimen of FLASH radiotherapy and followed post-treatment until subject death or lost to follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patient age at least 18 years
* 1 to 3 painful bone metastasis(-es) requiring treatment, in the ribs, clavicles, scapulae, or sternum (if more than one metastasis can be treated within the same treatment field, it will be counted as one metastatic site for the purpose of trial treatment).
* Bone metastases that can be treated within a field size up to 7.5 cm x 30 cm without overlap of radiation fields
* Life expectancy >6 months (in the judgement of the investigator)
* Patients who are able to comply with the protocol
* Provision of signed and dated informed consent form
* Clinically acceptable treatment plan

Exclusion Criteria:

* More than 3 painful bone metastases of the thorax requiring palliative radiotherapy (if more than one metastasis can be treated within the same treatment field, it will be counted as one metastatic site for the purpose of trial treatment).
* Overlap of FLASH radiation fields with any previous or planned radiation fields to the same site
* Patients with pathologic bone fractures in the treatment field
* Patients with metal implants in the treatment field
* Patients with symptomatic pneumonitis at the time of screening, or a history of symptomatic radiation pneumonitis
* Patients with known contraindications to thoracic radiation
* Patients who received or will receive cytotoxic chemotherapy and/or any prescribed systemic therapy known to impact tissue response to radiation, within 2 weeks prior or 1 week following their planned radiation treatment
* Prior local therapy modality to the treatment site(s) within 2 weeks of study enrollment that, in the judgement of the investigator, might compromise interpretation of pain response
* Patients with persistent toxicity > Grade 1 from prior systemic therapy within the proposed treatment field (with the exception of alopecia and peripheral neuropathy)
* Patients with pacemakers or other implanted devices at risk of malfunction during radiotherapy
* Patients with any other medical condition or laboratory value that would, at the discretion of the investigator, preclude the patient from participation in this clinical investigation
* Patients at known risk of enhanced normal tissue sensitivity to radiotherapy due to inherited predisposition or documented comorbidity that might lead to hypersensitivity to ionizing radiation
* Patients enrolled in any other clinical studies that the investigator believes to be in conflict with this clinical investigation.
* Patients who are pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-03-08 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of radiation-related toxicities that are possibly, probably, or definitely related to FLASH radiotherapy. | Assessed from start of treatment until 6 months post treatment.
  Toxicities that are possibly, probably, or definitely related to FLASH radiotherapy. Toxicities will be classified per CTCAE version 5.0.
Assessment of pain relief using patient reported pain questionnaire for overall pain score | Change from baseline pain overall at 3 months.
  Patient reported pain overall
Assessment of pain relief using patient reported pain questionnaire for pain at treated site | Change from baseline pain at treated site at 3 months.
  Patient reported pain at treated site
Use of pain medication | Change from baseline pain medication usage at 3 months.
  Capture dose and frequency of pain medication usage or pain medication changes.

SECONDARY OUTCOMES:
Workflow feasibility - time on table | Will be assessed on day of treatment delivery which occurs within 2-4 weeks of subject enrollment.
  Total subject treatment time on table.
Workflow feasibility - delays in study treatment | Will be assessed on day of treatment delivery which occurs within 2-4 weeks of subject enrollment.
  Treatment for an individual subject will be deemed NOT feasible if delays in study treatment of more than 10 business days from simulation to treatment occurs related to the investigational device (excluding delays due to patient or facility factors not related to study treatment).

CONTACTS AND LOCATIONS:
Overall Officials: John Perentesis, MD, Principal Investigator — Medical Director Cincinnati Children's/UC Health Proton Therapy Center
Locations (2):
- United States (2):
  - OSF Healthcare Saint Francis Medical Center, Peoria, Illinois
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Daugherty EC, Zhang Y, Xiao Z, Mascia AE, Sertorio M, Woo J, McCann C, Russell KJ, Sharma RA, Khuntia D, Bradley JD, Simone CB 2nd, Breneman JC, Perentesis JP. FLASH radiotherapy for the treatment of symptomatic bone metastases in the thorax (FAST-02): protocol for a prospective study of a novel radiotherapy approach. Radiat Oncol. 2024 Mar 12;19(1):34. doi: 10.1186/s13014-024-02419-4. PMID 38475815